CLINICAL TRIAL: NCT04337125
Title: Cross-sectional Study Assessing the Contribution of Attachment and Educational Practices in the Expression of ADHD in School-aged ADHD Children and Control Group
Brief Title: Contribution of Attachment and Educational Practices in the Expression of ADHD in School-aged Children
Acronym: CASPI-ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Fabiola Children's University Hospital (Other)
Collaborators: The Belgian Kids' Fund (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P2020/PSY/CASPI-ADHD
Record Dates: First submitted 2020-04-01; First posted 2020-04-07 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: child; attachment; parenting; ADHD; executive functions
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADHD group (Other): ADHD children with their parents
  Interventions: Other: Neuropsychological and attachment/parenting assessment
- Control group (Other): Children with typical development and their parents
  Interventions: Other: Neuropsychological and attachment/parenting assessment

INTERVENTIONS:
Other: Neuropsychological and attachment/parenting assessment — Children assessments:
  Mental health assessment, Intellectual functioning assessment, Sleep patterns assessment, Behavior assessment, Severity of ADHD symptoms assessment, child attachment assessment, parenting practices assessment, emotional regulation assessment, Direct measures of attention and executive functions assessment, Indirect measures of attention and executive functions assessment
  Parents assessments:
  Mental health assessment, Intellectual functioning assessment, ADHD symptoms assessment, Depression symptoms assessment, Attachment style assessment, Direct measures of attention and executive functions assessment, Indirect measures of attention and executive functions assessment.

SUMMARY:
ADHD is a neurodevelopmental disorder characterized by the presence of persistent signs of associated hyperactivity-impulsivity and/or inattention that impair the child's functioning or development.

The involvement of genetic factors has been shown in numerous studies. Other studies have also highlighted the contributions of parent-child interaction in the development, expression and persistence of symptoms.However, the mechanisms by which parenting practices and attachment may influence ADHD symptoms remain unclear.

The aim of this study is to evaluate the influence of attachment style of the child, the educational practices and the presence of attentional/executive disorders of parents on the expression of ADHD in children aged 7 to 10.

This prospective empirical research will compare children with ADHD and their parents to a matched control group.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients ages 7 to ≤10 years with ADHD (study group) or TD children matched by gender and socio-economic factors (control group) and their parents.

French-speaking population Willing and able to comply with scheduled visits and study procedures. Written informed consent/assent, according to local guidelines, signed by the patient and / or by the parents or legal guardian prior to any study related screening procedures are performed.

Exclusion Criteria:

Children with intellectual disabilities (IQ <80). Epilepsy. Prematurity. Objectified neurological sequelae. Specific language impairment or severe learning disabilities. Contraindication to stopping treatment for ADHD

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cartes pour l'évaluation de l'Attachement et de la Mentalisation chez l'Enfant (CAME) | At enrollment
  CAME is a child interview validated in french and allowing to assess the attachment representations and mentalization on base of interview for child between 7 and 14 years. The aim of interview is to tell the child the emotional relationships with parents (e.g. : "Can you tell me a moment where your mom/dad was mad at you" ? or "did you ever feel bad about yourself, feel bad about yourself ? "). The interview with child is recorded and transcribed word for word for the correction. In order to increasing quality of rating, 20% of interview will be recorded by a second evaluator (Pr Ayala Borghini)
Security Scale - version français (SS-vf) | At enrollment
  The child is asked to complete two questionnaires with each 10 items, one for the mother, the other for the father. Responses to each item are scored on a 4-point scale. In the version validated in French, the scores vary from 10 to 40. The highest scores correspond to the highest security of attachment to the parent.

SECONDARY OUTCOMES:
Parent Education Practices Assessment Questionnaire (PEP) | At enrollment
  PEP is a questionaire completed by parents to assess parents' child-rearing behavior and included 35 questions divided into 9 factors: positive parenting, monitoring, rules, punishment, ignorance, maternal reward and autonomy.
  This questionnaire will be used to compare the distribution of parenting practices in children with AHDH and with TD group
Parent Educational Practices perceived by the child (PEPPE) | At enrollment
  PEPPE is a questionaire completed by child and is composed to 18 questions to assess perception of parenting practices.
Behavioral Rating Inventory Executive Function (BRIEF) | At enrollment
  BRIEF is a questionnaire rated by parents to assess child's executive functioning and is composed of a 86 items. Each item is rated on 0-2 scale. Higher scores indicate more executive difficulties.
Behavioral Rating Inventory Executive Function for Adult (BRIEF-A) | At enrollment
  BRIEF-A is a self-report to assess parent's executive functioning in parent and includes 75 items. Each item is rated on 0-2 scale. Higher scores indicate more executive difficulties.
Test of Attentional Performance (TAP) | At enrollment
  TAP is a computerized battery allowing attentional performances and different executive functions such as alertness, divided attention, motor inhibition, flexibility.
Stroop | At enrollment
  This task includes three conditions: denomination, reading, interference. In the denomination condition, adult must saw as quickly as possible the color of each square presented in line. In the reading condition adult must read as quickly as the name of colors presented in line in black ink (congruent condition). In the interference condition, he must say the color of the ink of word (names of colors in a different ink than the color named) and thus inhibit the automatic treatment of read.
Counting Stroop Task | At enrollment
  This task includes three conditions : counting, reading, interference. Items were presented on a computer screen in 10 lines, presented one at time, with 10 stimuli per line (squares with numbers or dots). In the counting condition, children had to report as fast as possible the number of dots within each square. In the reading condition, they had to read the number written within each square. In the interference condition, they had to report how many numbers were written within each square, while avoiding reading the number itself. Important variables for analysis are number of errors and time in interference condition.
Tower of London | At enrollment
  The test consists of a support with three rods of different heights and three beads of different colors. The individual must reproduce, on the support and in a determined number of movements, a particular configuration proposed by the examiner. Important variable is the number of excess movements.
Attention Deficit Hyperactivity Disorder-Rating Scale (ADHD-RS) | At enrollment
  ADHD-RS is a questionnaire rated by parents to assess severity of ADHD and is composed of 18 items on 0-3 point scale. Higher scores indicates more ADHD symptoms.
Emotional Regulation Checklist - version française (ERC-vf) | At enrollment
  ERC-vf is a questionnaire rated by parents to assess abilities of emotional regulation and emotional dysregulation of child and is composed to 24 items divided in two scale. Each item is rated on 0-4 scale. Higher score in emotional dysregulation scale indicate more difficulty. Higher score in scale of emotional regulation indicate more competence for regulate emotions.
Children Behavior Checklist (CBCL) | At enrollment
  CBCL is a questionnaire rated by parents to assess child's behavior and presence of comorbid disorders such as anxiety, depression or oppositional disorders and is composed of 118 items. Each item is rated on 0-2 scale. Raw scores were converted on T-scores on three large scales (Internalising, Externalising, Total) and eight syndrome scales (Aggressive Behavior, Anxious/Depressed, Attention, Problems, Rule-Breaking Behavior, Social Problems, Somatic Complaints, Thought Problems, Withdrawn/Depressed). Higher scores indicate more difficulty.
Revised Card Sorting Test (RCST) | At enrollment
  Cognitive flexibility of child will be assessed with RCST. Children must classed a set of 48 card according to three possibles categories (color, shape and number). Child must inferred the correct category on base examinator feedback. Important variable is the number of errors.
Kiddie-SADS-PL | At enrollment
  The evaluation of child and adolescent mental health disorder is assessed by the Kiddie-SADS-PL DSM-5, a semi-structured diagnostic interview for children and adolescents
Wechsler Intelligence Scale for Children 5th edition (WISC-V) | At enrollment
  The child intellectual functioning will be assessed using the WISC-V (Wechsler, 2016). The Digit span subtest will be using as measure of working memory
Wechsler Adult Intelligence Scale 4th edition (WAIS-IV) | At enrollment
  The parental intellectual functioning will be assessed with the WAIS-IV subtests of Matrices and Figure weight. The Digit span subtest will be using as measure of working memory.
Mini International Neuropsychiatric Interview (MINI) | At enrollment
  MINI is a semi-structured diagnostic interview for adults validated in french (Lecrubier & al., 1997). Current and past symptoms of psychopathology are assessed in order to establish one or more diagnoses according to the DSM-5 criteria.
ADHD Adult Scale Rating Scale (ASRS) | At enrollment
  ASRS is a self-questionnaire to assess presence and severity of ADHD symptoms in parents and is composed of 18 items on 0-3 point scale. Higher scores indicates more ADHD symptoms.
Wenders Utah Rating Scale (WURS) | At enrollment
  WURS is a self-questionnaire completed by parent that allows to assess retrospectively the presence of attentional difficulties and hyperactivity signs in childhood. The french version included 25 items rated from 0 to 4 depending on the severity of the behavior. Higher scores indicate more difficulty.
Relationship Scale Questionnaire (RSQ) | At enrollment
  RSQ is a self-questionnaire of 30 items destined to assess the attachment style of adult (Secure, Fearful, Preoccupied and Detached). The adult rates each item on Likert scale in 5 points according to what looks most like him.
Beck Depression Inventory-II (BDI-II) | At enrollment
  BDI-II is a self-report to assess presence of depressive symptoms in parent and includes 21 items. Each item is rated on 0-3 scale. Higher scores indicate more depressive symptoms
Children's Sleep Habit Questionnaire (CSHQ) | At enrollment
  CSHQ is questionnaire rated by parents and is composed of 35 items on 1-3 point scale. Higher scores indicates more sleep disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Delvenne, MDPhD, Study Director — Queen Fabiola Children's University Hospital
Locations (2):
- Belgium (2):
  - Hôpital Universitaire Des Enfants Reine Fabiola, Brussels
  - Hôpital Erasme, Brussels

IPD SHARING:
Plan to Share IPD: No